CLINICAL TRIAL: NCT06114056
Title: A Clinical Study Evaluating the Safety, Tolerability, and Initial Efficacy of Single Intravenous Infusion of JWK007 in Patients With Duchenne Muscular Dystrophy (DMD)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1285
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Gene Therapy; Adeno-associated virus
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JWK007 injection (Experimental): AAVrh74 was used as the vector for JWK007 injection. Because the Dystrophin gene is too large to be used for conventional rAAV loading (AAV packaging capacity < 5.0kb), we independently designed a new micro-dystrophin (μDystrophin) for each functional domain of the gene. The protein includes structures essential for promoting neuronal nitric oxide synthase (nNOS) activity and membrane-binding domains.
  Interventions: Biological: JWK007 Single intravenous infusion administration

INTERVENTIONS:
Biological: JWK007 Single intravenous infusion administration — Six male children aged 5-10 years were enrolled in the study. The patients were divided into two different dose groups, and a "3+3" dose escalation design was used, the low dose was 1.0×1014vg/kg, and the high dose was 2.0×1014vg/kg. Only one intravenous infusion of JWK007 was administered to each patient.

SUMMARY:
This study is a single-center, single-arm, non-randomized, open-label, non-controlled, dose-escalation, prospective clinical trial designed to assess the safety, tolerability, and preliminary efficacy of JWK007 injection in pediatric patients with Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
DMD is a rare genetic disorder that primarily affects males. This disease is closely associated with mutations in the DMD gene located on the X chromosome. The DMD gene encodes a protein known as dystrophin, which plays a crucial role in providing essential structural and protective support within the muscles. Gene therapy drugs using Adeno-Associated Virus (AAV) as a vector hold the promise of offering a convenient, effective, and safe treatment option for DMD patients. Therefore, we have independently developed and designed the JWK007 injection. The study will include two dosing groups and employ a '3+3' dose escalation design, incrementally increasing dosages in a sequential, ascending manner.

ELIGIBILITY:
Inclusion Criteria:

Participants meeting all of the following criteria may be considered for inclusion:

1. Male, aged 5 to 10 years (inclusive).
2. Diagnosis of Duchenne Muscular Dystrophy (DMD) confirmed through medical history and genetic testing, characterized by a frameshift mutation (deletion or duplication) or a premature stop codon mutation in the DMD gene between exons 18 to 58.
3. Below-average performance on motor assessment testing.
4. Ability to cooperate with motor assessment testing.
5. Tolerance for muscle biopsy under anesthesia with no contraindications for biopsy.
6. Participants must have been taking a stable dose of oral corticosteroids for at least 12 weeks prior to screening, and the expected dose should remain constant throughout the study, except for adjustments related to changes in body weight.

Exclusion Criteria:

Participants meeting any one of the following criteria are not eligible for inclusion:

1. Active viral infection based on clinical observations.
2. Signs of cardiomyopathy, including echocardiogram with ejection fraction below 40%.
3. Serological evidence of HIV infection, or Hepatitis B or C infection.
4. Diagnosis of (or ongoing treatment for) an autoimmune disease.
5. Abnormal laboratory values considered clinically significant (GGT > 3XULN, bilirubin ≥ 3.0 mg/dL, creatinine ≥ 1.8 mg/dL, Hgb < 80 or > 180 g/L; WBC > 18.5*10^9/L).
6. Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer.
7. Subjects with AAVrh74 neutralizing antibody titers > 1:400 as determined by ELISA immunoassay.
8. Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's wellbeing, safety, or clinical interpretability.
9. Severe infection (eg. pneumonia, pyelonephritis, or meningitis) within 4 weeks before gene transfer visit (enrollment may be postponed).
10. Has received any investigational medication (other than corticosteroids) or exon skipping medications (including ExonDys 51), experimental or otherwise, in the last 6 months prior to screening for this study.
11. Has had any type of gene therapy, cell based therapy (eg. stem cell transplantation), or CRISPR/Cas9.
12. Family does not want to disclose patient's study participation with primary care physician and other medical providers

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2029-11-13 (Estimated); Study Completion 2029-11-13 (Estimated)

PRIMARY OUTCOMES:
adverse events | 5 years
  Adverse events defined as the number of participants with adverse events according CTCAE v5.0

SECONDARY OUTCOMES:
North Star Ambulatory Assessment | 5 years
  North Star Ambulatory Assessment (NSAA) is a clinical tool used to assess the motor function and ambulatory capabilities of children and adolescents with neuromuscular disorders like Duchenne muscular dystrophy.
Six-Minute Walk Test | 5 years
  the distance the patient walked in six minutes
10-Meter Walk/Run Test | 5 years
  The time it takes to walk 100 meters
creatine kinase | 5 years
  Changes in circulating levels of CK
the expression of micro-dystrophin gene | 6 months
  Baseline muscle biopsies for dystrophin expression will be performed between -30 and -7 days prior to treatment in all subjects. All subjects will undergo a post-treatment biopsy on day 180. Micro-dystrophin gene expression was quantified (immunofluorescence and Western blot analysis) and compared before and after muscle biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Xingchen, Ph.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa Verdera H, Kuranda K, Mingozzi F. AAV Vector Immunogenicity in Humans: A Long Journey to Successful Gene Transfer. Mol Ther. 2020 Mar 4;28(3):723-746. doi: 10.1016/j.ymthe.2019.12.010. Epub 2020 Jan 10. PMID 31972133
- [Background] Mendell JR, Sahenk Z, Lehman K, Nease C, Lowes LP, Miller NF, Iammarino MA, Alfano LN, Nicholl A, Al-Zaidy S, Lewis S, Church K, Shell R, Cripe LH, Potter RA, Griffin DA, Pozsgai E, Dugar A, Hogan M, Rodino-Klapac LR. Assessment of Systemic Delivery of rAAVrh74.MHCK7.micro-dystrophin in Children With Duchenne Muscular Dystrophy: A Nonrandomized Controlled Trial. JAMA Neurol. 2020 Sep 1;77(9):1122-1131. doi: 10.1001/jamaneurol.2020.1484. PMID 32539076
- [Background] Miesbach W, Meijer K, Coppens M, Kampmann P, Klamroth R, Schutgens R, Tangelder M, Castaman G, Schwable J, Bonig H, Seifried E, Cattaneo F, Meyer C, Leebeek FWG. Gene therapy with adeno-associated virus vector 5-human factor IX in adults with hemophilia B. Blood. 2018 Mar 1;131(9):1022-1031. doi: 10.1182/blood-2017-09-804419. Epub 2017 Dec 15. PMID 29246900
- [Background] Duan D. Systemic AAV Micro-dystrophin Gene Therapy for Duchenne Muscular Dystrophy. Mol Ther. 2018 Oct 3;26(10):2337-2356. doi: 10.1016/j.ymthe.2018.07.011. Epub 2018 Jul 17. PMID 30093306
- [Background] Xue F, Li H, Wu X, Liu W, Zhang F, Tang D, Chen Y, Wang W, Chi Y, Zheng J, Du Z, Jiang W, Zhong C, Wei J, Zhu P, Fu R, Liu X, Chen L, Pei X, Sun J, Cheng T, Yang R, Xiao X, Zhang L. Safety and activity of an engineered, liver-tropic adeno-associated virus vector expressing a hyperactive Padua factor IX administered with prophylactic glucocorticoids in patients with haemophilia B: a single-centre, single-arm, phase 1, pilot trial. Lancet Haematol. 2022 Jul;9(7):e504-e513. doi: 10.1016/S2352-3026(22)00113-2. Epub 2022 May 19. PMID 35598604
- [Background] Roberts TC, Wood MJA, Davies KE. Therapeutic approaches for Duchenne muscular dystrophy. Nat Rev Drug Discov. 2023 Nov;22(11):917-934. doi: 10.1038/s41573-023-00775-6. Epub 2023 Aug 31. PMID 37652974